CLINICAL TRIAL: NCT06537531
Title: Video Classification of Intubation in Spain
Brief Title: Video Classification of Intubation in Spain (VCI)
Acronym: VCI
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: 2022.079
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Difficult Intubation
Keywords: Difficult intubation; Airway; Videolaryngoscopy; Score

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients from any geographical area of the Iberian Peninsula who decide to undergo scheduled surgery at our hospital during a period of 6 months (2024-25).
  Interventions: Other: Compare VCI scale

INTERVENTIONS:
Other: Compare VCI scale — Compare VCI scale

SUMMARY:
Use of VCI in Spain

DETAILED DESCRIPTION:
The clinical importance of airway management has gained relevance over the last decade in most scientific societies with the objective of improving the standard of care.

The WHO has focused its guidelines on "Safe Surgery," aiming to encompass all methods that predict and recognize the risk of difficult airway management or aspiration, which must be applied by the surgical team. To this end, it has created and implemented a surgical safety checklist that can be useful in reducing the risk of unidentified difficulties.

The same suggestion has been included in the Helsinki Declaration on Patient Safety in Anesthesiology, endorsed by most European entities in cooperation with the European Society of Anesthesiology (ESA), the European Board of Anesthesiology (EBA-UEMS), the World Federation of Societies of Anesthesiology (WFA), and the European Patients' Federation (EPF). The protocol for difficult airway management and the implications of the Helsinki Declaration were published in 2013 in the Spanish Journal of Anesthesiology and Resuscitation.

Airway management today is perhaps the field that most concerns anesthesiologists, as decisions and actions must be taken quickly and effectively when facing a potential difficult airway (DA). Failure to do so would result in significant morbidity and mortality for patients.

The incidence of difficulty in orotracheal intubation (OTI) ranges between 1.5% and 13%. Most errors in airway management are due to ignorance and the low reliability of traditional protocols, algorithms, and combinations of detection tools to identify a potentially difficult airway.

This field is constantly evolving, and in the last 20 years, we have witnessed the emergence of a large number of devices: Supraglottic Devices (SGDs) or Extraglottic Devices (EGDs) in the past decade, and Optical Devices (videolaryngoscopes) in this last decade.

The existence of a large number of new devices in this field implies a deep understanding of these, both theoretically and practically, during scheduled surgery. Once this is achieved, practitioners should know how to use them appropriately in DA situations.

Since 1993, when the American Society of Anesthesiology (ASA) published its "Recommendations for Difficult Airway Management," many countries and scientific societies have created their protocols, guidelines, and algorithms that we must know and apply, always adapting them to our environment and the available devices.

In Spain, since the mid-1990s, DA training programs for specialist doctors have been launched, gradually expanding and covering all personnel involved in airway management. Today, training in this field has become part of the knowledge and skills acquisition in various specialties, notably Anesthesiology and Resuscitation.

The phrase "prevention is better than cure" is an intuitive, acceptable, and politically correct concept. This is applicable in our field since, although there are not many patient factors we can modify (anatomy is intrinsic), there are possible modifications in our actions that can determine the success or failure in airway management.

Currently, there is no universally accepted method for describing tracheal intubation via videolaryngoscopy. It is important that this information is communicated and documented accurately to plan airway management procedures for the patient, thereby improving care safety. The Intubation Classification Scale or Video Intubation Classification (VCI) score has been proposed to succinctly describe the key practical elements of tracheal intubation via videolaryngoscopy in the order they are performed. This classification consists of three sections: the first describes the type of blade used (Macintosh or hyperangulated), the second describes the POGO (Percentage of Glottic Opening) at the time of intubation, and finally, the ease/difficulty or impossibility of inserting the tube through the glottis.

ELIGIBILITY:
Inclusion Criteria:

* Patients from any geographical area of the Iberian Peninsula who decide to undergo scheduled surgery at our hospital during a period of 6 months (2024-25).

Exclusion Criteria:

* Age <18

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from any geographical area of the Iberian Peninsula who decide to undergo scheduled surgery at our hospital during a period of 6 months (2024-25).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
VCI scale from observer (1-4) | 2 minutes
  VCI scale from observer(1-4)
VCI scale from intubator (1-4) | 2 minutes
  VCI scale from intubator (1-4)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clinica Universidad de Navarra, Madrid, Madrid
  - Miguel Angel Fernandez-Vaquero, Madrid, Madrid

REFERENCES:
- [Derived] Fernandez-Vaquero MA, Charco-Mora P, Sastre-Rincon JA, Gomez-Rios MA, Cardenas-Gomez J, Martinez-Hurtado E, Aracil-Escoda N, Vallejo-Tarrat A, Thion-Soriano I, Peral-Sanchez D, Castaneda-Pascual M, Rodriguez Del Rio M, de Luis-Cabezon N, Gonzalez-Garcia J, Acosta-Martinez J, Gonzalez-Santos S, Onrubia-Fuertes X, Martinez-Gonzalez E, Roca de Togores-Lopez A, Gonzalez-Mendibil I, Banos-Maestro A, Mariscal-Flores M, Lluch-Oltra A, Emazabel-Yunta I, Rodriguez-Sanabria DM, Alvarez-Avello JM, Melendez Salinas DA, Lopez-Correa T, Sanchez-Merchante M, Bermudez-Lopez M, Martinez-Gallego E, Martinez-Segovia MC, Martin-Andres AB, Molero-Diez Y, Garcia-Aroca MA, Tapia-Salinas B, Puig-Bernabe J, Piano A, Hernandez-Fernandez G, Mingote-Llado A, Garcia-Fernandez J, Mata-Estevez J, Reviriego-Agudo L, Ruiz-Cordoba G, Moya-Moradas J, Marques-Asin FJ, Santacana MV; VCISpain Trial Investigators Group. VCISpain: protocol for a prospective multicenter observational study to validate a standardized classification tool for tracheal intubation using videolaryngoscopy. Braz J Anesthesiol. 2025 Sep-Oct;75(5):844653. doi: 10.1016/j.bjane.2025.844653. Epub 2025 Jun 18. PMID 40553732